CLINICAL TRIAL: NCT03875482
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of Risankizumab Using a New Formulation for the Treatment of Adult Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Assess Safety and Efficacy of Risankizumab Using a New Formulation in Participants With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-999
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Psoriasis
Keywords: Risankizumab; Psoriasis; Plaque Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Risankizumab (Experimental): Subcutaneous (SC), self-administered 150 mg doses of risankizumab at Weeks 0, 4, and 16
  Interventions: Drug: Risankizumab
- Placebo (Placebo Comparator): Subcutaneous (SC), self-administered doses of placebo solution at Weeks 0, 4, and 16
  Interventions: Drug: Placebo solution for risankizumab

INTERVENTIONS:
Drug: Risankizumab — Risankizumab 150 mg (150 mg/mL) in prefilled syringes, self-administered subcutaneously
  Other Names: ABBV-066; BI 655066
  Arms: Risankizumab
Drug: Placebo solution for risankizumab — Placebo solution in prefilled syringes, self-administered subcutaneously
  Arms: Placebo

SUMMARY:
The primary objective of this study was to evaluate the safety and efficacy of risankizumab (150 mg/mL) administered by prefilled syringe (PFS) for the treatment of adult participants with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This was a Phase 3, multicenter, randomized, double-blind, placebo-controlled, parallel group study to evaluate the safety and efficacy of risankizumab 150 mg/mL formulation in PFS in adult participants with moderate to severe plaque psoriasis. The study included a 30-day screening period, a 28-week treatment period with study visits at Weeks 0, 4, 16 and 28, and a subsequent follow-up telephone call at approximately 20 weeks after the last dose of study drug. Study drug dosing consisted of 3 self-administered, subcutaneous (SC) doses on Weeks 0, 4, and 16. Dosing on Week 4 was self-administered at home.

ELIGIBILITY:
Inclusion Criteria:

* Participant has diagnosis of chronic plaque psoriasis for at least 6 months before the baseline visit.
* Participant meets following disease activity criteria:
* Stable moderate to severe chronic plaque psoriasis, defined as greater than or equal to 10% body surface area (BSA) psoriasis involvement, static physician global assessment (sPGA) score of greater than or equal to 3, and Psoriasis Area Severity Index (PASI) greater than or equal to 12 at Screening and baseline visit.
* Candidate for systemic therapy as assessed by the investigator.

Exclusion Criteria:

* Participant has history of active skin disease other than psoriasis that could interfere with the assessment of psoriasis.
* Participant has history of erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis.
* Participant has previous exposure to risankizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (43):
- United States (40):
  - Total Skin and Beauty Derm Ctr /ID# 210366, Birmingham, Alabama
  - Alliance Dermatology and MOHs /ID# 210645, Phoenix, Arizona
  - Hull Dermatology, PA /ID# 210305, Rogers, Arkansas
  - Anaheim Clinical Trials LLC /ID# 212559, Anaheim, California
  - Wallace Medical Group, Inc. /ID# 210403, Beverly Hills, California
  - Dermatology Res. Assoc., CA /ID# 210402, Los Angeles, California
  - Integrative Skin Science and Research /ID# 212551, Sacramento, California
  - Mosaic Dermatology /ID# 210780, Santa Monica, California
  - Skin Care Research, LLC /ID# 210514, Boca Raton, Florida
  - ACCEL Research Sites /ID# 212709, DeLand, Florida
  - Multi-Speciality Research Associates /ID# 211625, Lake City, Florida
  - GSI Clinical Research, LLC /ID# 210330, Margate, Florida
  - Suncoast Clinical Research /ID# 210874, New Port Richey, Florida
  - Ormond Medical Arts Pharmaceutical Research Center /ID# 212781, Ormond Beach, Florida
  - Progressive Medical Research /ID# 210877, Port Orange, Florida
  - Precision Clinical Research /ID# 212921, Sunrise, Florida
  - Lenus Research & Medical Group /ID# 212584, Sweetwater, Florida
  - Treasure Valley Dermatology /ID# 212707, Boise, Idaho
  - Sneeze, Wheeze, & Itch Associates, LLC /ID# 212562, Normal, Illinois
  - The Indiana Clinical Trials Center /ID# 210205, Plainfield, Indiana
  - Forefront Dermatology /ID# 210520, Louisville, Kentucky
  - DS Research /ID# 210272, Louisville, Kentucky
  - David Fivenson, MD, PLC /ID# 210193, Ann Arbor, Michigan
  - Clarkston Skin Research /ID# 210197, Clarkston, Michigan
  - Henry Ford Medical Center /ID# 211598, Detroit, Michigan
  - Cleaver Dermatology /ID# 210300, Kirksville, Missouri
  - Advanced Dermatology of the Midlands /ID# 212763, Omaha, Nebraska
  - Skin Specialists, PC /ID# 211490, Omaha, Nebraska
  - Psoriasis Treatment Ctr NJ /ID# 210837, East Windsor, New Jersey
  - Skin Laser and Surgery Specialists of NY and NJ /ID# 210208, Hackensack, New Jersey
  - DermResearchCenter of NY, Inc. /ID# 210652, Stony Brook, New York
  - WDC Cosmetic and Research, PLLC /ID# 210372, Wilmington, North Carolina
  - Lynn Health Science Institute (LHSI) /ID# 213216, Oklahoma City, Oklahoma
  - Clinical Partners, LLC /ID# 210642, Johnston, Rhode Island
  - Palmetto Clinical Trial Services /ID# 210368, Fountain Inn, South Carolina
  - Coastal Carolina Research Ctr /ID# 213069, Mt. Pleasant, South Carolina
  - Arlington Research Center, Inc /ID# 210344, Arlington, Texas
  - Center for Clinical Studies - Houston (Binz) /ID# 210361, Houston, Texas
  - Progressive Clinical Research /ID# 210359, San Antonio, Texas
  - Acclaim Dermatology /ID# 212252, Sugar Land, Texas
- Puerto Rico (3):
  - Dr. Samuel Sanchez, PSC /ID# 211142, Caguas
  - Pan American Center for Oncology Trials, LLC /ID# 212445, Rio Piedras
  - Clinical Research Puerto Rico /ID# 211144, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Blauvelt A, Gordon KB, Lee P, Bagel J, Sofen H, Lockshin B, Soliman AM, Geng Z, Zhan T, Alperovich G, Stein Gold L. Efficacy, safety, usability, and acceptability of risankizumab 150 mg formulation administered by prefilled syringe or by an autoinjector for moderate to severe plaque psoriasis. J Dermatolog Treat. 2022 Jun;33(4):2085-2093. doi: 10.1080/09546634.2021.1914812. Epub 2021 May 5. PMID 33947295
- See also: Related Info. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intent-to-treat (ITT) population: all randomized participants
Period: Overall Study
Arm/Group | Risankizumab | Placebo
Started | 105 | 52
Completed | 92 | 32
Not Completed | 13 | 20
Not completed — Adverse Event | 0 | 1
Not completed — Withdrew consent | 5 | 6
Not completed — Lost to Follow-up | 8 | 2
Not completed — Lack of Efficacy | 0 | 11

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Risankizumab | Placebo | Total
Number analyzed (Participants) | 105 | 52 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (15.14) | 48.8 (15.47) | 49.1 (15.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 24 | 70
  Male | 59 | 28 | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 87 | 44 | 131
  Black or African American | 12 | 4 | 16
  Asian | 3 | 1 | 4
  American Indian or Alaska Native | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 1 | 2 | 3
  Multiple | 1 | 1 | 2
Prior Use of Systemic Biologic for Psoriasis [Count of Participants; unit: Participants]
  0 | 58 | 29 | 87
  ≥1 | 47 | 23 | 70
Static Physician Global Assessment (sPGA) Score at Baseline [Count of Participants; unit: Participants] — The sPGA is an investigator assessment of the overall disease severity at the time of evaluation. Erythema, induration, and scaling of psoriatic lesions are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA ranges from 0 to 4, and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean >0, <1.5; Mild (2) = mean ≥1.5, <2.5; Moderate (3) = mean ≥2.5, <3.5; and Severe (4) = mean ≥3.5.
  Participants
    Score of 3 | 86 | 46 | 132
    Score of 4 | 19 | 6 | 25
Psoriasis Area and Severity Index (PASI) Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — The PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.
  units on a scale | 21.529 (9.5975) | 21.060 (10.2563) | 21.373 (9.7901)
Body Surface Area (BSA) Psoriasis Involvement at Baseline [Mean (Standard Deviation); unit: Percentage of body surface area affected] | 28.343 (16.4139) | 28.160 (18.4868) | 28.282 (17.0689)
Duration of Plaque Psoriasis [Mean (Standard Deviation); unit: years] | 20.91 (13.837) | 15.82 (11.753) | 19.22 (13.363)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Psoriasis Area Severity Index (PASI) 90 at Week 16
Description: The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at Week 16) / PASI score at Baseline * 100.
Time Frame: At Week 16
Population: Intent-to-treat (ITT) population: all randomized participants; those with missing data were imputed as non-responders
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab | Placebo
Number analyzed (Participants) | 105 | 52
percentage of participants | 62.9 [53.6 to 72.1] | 3.8 [0.0 to 9.1]
Statistical Analysis 1: Comparison: Risankizumab vs Placebo; The variable was analyzed using the Chi-square test. Both null hypotheses corresponding to the co-primary endpoints must be rejected simultaneously under a two-sided significance level of 0.05; Test type: Superiority; p < 0.001, Chi-squared; Mean Difference = 59.0, 95% CI 2-sided [48.4 to 69.6]

2. Primary Outcome: Percentage of Participants Achieving Static Physician Global Assessment (sPGA) of Clear or Almost Clear at Week 16
Description: The sPGA is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema, induration, and scaling of psoriatic lesions are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA ranges from 0 to 4, and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean >0, <1.5; Mild (2) = mean ≥1.5, <2.5; Moderate (3) = mean ≥2.5, <3.5; and Severe (4) = mean ≥3.5.
Time Frame: At Week 16
Population: Intent-to-treat (ITT) population: all randomized participants; those with missing data were imputed as non-responders
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab | Placebo
Number analyzed (Participants) | 105 | 52
percentage of participants | 78.1 [70.2 to 86.0] | 9.6 [1.6 to 17.6]
Statistical Analysis 1: Comparison: Risankizumab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Chi-squared; Mean Difference = 68.5, 95% CI 2-sided [57.2 to 79.7]

3. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area Severity Index (PASI) 100 at Week 16
Description: The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI100 is defined as a 100% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at Week 16) / PASI score at Baseline * 100.
Time Frame: At Week 16
Population: Intent-to-treat (ITT) population: all randomized participants; those with missing data were imputed as non-responders
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab | Placebo
Number analyzed (Participants) | 105 | 52
percentage of participants | 38.1 [28.8 to 47.4] | 1.9 [0.0 to 5.7]
Statistical Analysis 1: Comparison: Risankizumab vs Placebo; The ranked secondary efficacy endpoints at Week 16 were to be tested between the risankizumab and placebo treatment groups among the ITT Population in a hierarchical order only if the null hypotheses for both primary endpoints had been rejected; Test type: Superiority; p < 0.001, Chi-squared; Mean Difference = 36.2, 95% CI 2-sided [26.2 to 46.2]

4. Secondary Outcome: Percentage of Participants Achieving Static Physician Global Assessment (sPGA) of Clear at Week 16
Description: as for outcome 2
Time Frame: At Week 16
Population: Intent-to-treat (ITT) population: all randomized participants; those with missing data were imputed as non-responders
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab | Placebo
Number analyzed (Participants) | 105 | 52
percentage of participants | 39.0 [29.7 to 48.4] | 1.9 [0.0 to 5.7]
Statistical Analysis 1: Comparison: Risankizumab vs Placebo; The ranked secondary efficacy endpoints at Week 16 were to be tested between the risankizumab and placebo treatment groups among the ITT Population in a hierarchical order only if the null hypotheses for both primary endpoints and for the first secondary endpoint had been rejected; Test type: Superiority; p < 0.001, Chi-squared; Mean Difference = 37.1, 95% CI 2-sided [27.1 to 47.2]

5. Other Pre Specified Outcome: Percent Change From Baseline in Psoriasis Area Severity Index (PASI) Score up to Week 16
Description: The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked.The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. Negative values indicate an improvement from baseline.
Time Frame: Baseline, Week 4, and Week 16
Population: Intent-to-treat (ITT) population: all randomized participants with a non-missing baseline measurement and at least one post-baseline value
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from Baseline
Arm/Group | Risankizumab | Placebo
Number analyzed (Participants) | 101 | 50
percent change from Baseline
  Week 4 | -50.62 [-56.255 to -44.987] | -14.48 [-22.490 to -6.470]
  Week 16: number analyzed (Participants) | 98 | 43
  Week 16 | -89.36 [-95.200 to -83.522] | -29.39 [-38.152 to -20.630]
Statistical Analysis 1: Comparison: Risankizumab vs Placebo; Risankizumab vs placebo at Week 4 Mixed-effect Model Repeat Measurements (MMRM): The repeated measures analysis was conducted using a mixed model including the baseline value and observed measurements at all post-baseline visits. The mixed model included the categorical fixed effects of treatment, visit and treatment-by-visit interaction as covariates; Test type: Superiority; p < 0.001, Mixed-effect Model Repeat Measurements; LS Mean Difference = -36.14, 95% CI 2-sided [-45.936 to -26.346], Standard Error of Mean 4.956 — Risankizumab - placebo
Statistical Analysis 2: Comparison: Risankizumab vs Placebo; Risankizumab vs placebo at Week 16 Mixed-effect Model Repeat Measurements (MMRM): The repeated measures analysis was conducted using a mixed model including the baseline value and observed measurements at all post-baseline visits. The mixed model included the categorical fixed effects of treatment, visit and treatment-by-visit interaction as covariates; Test type: Superiority; p < 0.001, Mixed-effect Model Repeat Measurements; LS Mean Difference = -59.97, 95% CI 2-sided [-70.501 to -49.439], Standard Error of Mean 5.326 — Risankizumab - placebo

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 20 weeks following discontinuation of study drug administration have elapsed, up to 48 weeks. In addition, serious adverse events were collected from the time the participant signed the study-specific informed consent.
Description: TEAEs and SAEs are defined as any AE or SAE with onset or worsening reported by a participant from the time that the first dose of study is administered until 20 weeks have elapsed following discontinuation of study drug. TEAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Risankizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/105 | 0/52
Other Adverse Events (participants affected / at risk) | 0/105 | 0/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risankizumab (N=105) | Placebo (N=52)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT03875482/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT03875482/SAP_001.pdf